CLINICAL TRIAL: NCT04769570
Title: Effect of Interscalene and Suprascapular Nerve Block on Analgesia Consumption After Adhesive Capsulitis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sibel Seçkin Pehlivan, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/580
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Shoulder Surgery
Keywords: suprascapular nerve block; interscalene brachial plexus block; ultrasound; patient satisfaction score; analgesic consumption
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group IPSB (Active Comparator): In the first group of patients (Group IPSB), ultrasound-guided interscalene brachial plexus block will be applied 30 minutes before surgery.
  Interventions: Procedure: interscalene brachial plexus block
- Group SSNB (Active Comparator): In the second group of patients, ultrasound-guided interscalene brachial plexus block and suprascapular nerve block will be applied 30 minutes before surgery.
  Interventions: Procedure: suprascapular nerve block
- Group Control (Active Comparator): Patients in the third group (Group C), will be considered the control group and no block will be performed.
  Interventions: Procedure: Group Control

INTERVENTIONS:
Procedure: interscalene brachial plexus block — Single shot ultrasound guided interscalene brachial plexus block will be performed preoperatively to patients.Patient-controlled analgesia (PCA) with morphine will be used for postoperative analgesia.
  Arms: Group IPSB
Procedure: suprascapular nerve block — Single shot ultrasound guided interscalene brachial plexus block and Suprascapular nerve block will be performed preoperatively to patients.Patient-controlled analgesia (PCA) with morphine will be used for postoperative analgesia.
  Arms: Group SSNB
Procedure: Group Control — consist of the patient group without any procedure.
  Arms: Group Control

SUMMARY:
In this study, a combination of different types of blocks for adhesive capsulitis surgery, the investigators will investigate the impact on patient satisfaction and analgesic consumption after surgery.

DETAILED DESCRIPTION:
General anesthesia will be performed in all patients for arthroscopic adhesive capsulitis shoulder surgeries. In the first group of patients (Group IPSB), interscalene brachial plexus block will be applied 30 minutes before surgery, while interscalene brachial plexus block and suprascapular nerve block (SSNB) administration to the second group patients (Group SSNB) before surgery. Patients in the third group (Group C) will be considered the control group and no block will be performed. Patient-controlled analgesia (PCA) with morphine will be used in all three groups for postoperative analgesia. Preoperative hemodynamic data of patients, postoperative pain scores (VAS), morphine consumption, patient satisfaction score, requirement of additional analgesia and observed side effects were recorded. Consumption of analgesia 24 hours after surgery and patient satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ASA I- ASA II Patients

Exclusion Criteria:

* history of allergy to the study medication
* refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Verbal Analogue Scores | 24 hours after surgery
  A research assistant, blinded to the group allocation, interviewed patients and collected data in the 24 hours postoperative period.Verbal Analog Pain Score value will be the lowest 0 and the highest 10. At the highest value, the patient's pain is at its maximum. and whether higher scores mean worse outcome.
opioid consumption | 24 hours after surgery
  In the recovery room all patients will be given a patient-controlled analgesia device containing morphine and 24 hours postoperative period will be recorded.

SECONDARY OUTCOMES:
Complications of the procedures | During the blocks and 24 hours after surgery
  The complications of the intervations will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Pehlivan, MD, Principal Investigator — TC Erciyes University
Locations (1):
- Sibel Seçkin Pehlivan, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De- identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 24 months of study completion.
Access Criteria: Data accept requests will be reviewed by an external independent Review Panel.

REFERENCES:
- [Result] Bowens C Jr, Sripada R. Regional blockade of the shoulder: approaches and outcomes. Anesthesiol Res Pract. 2012;2012:971963. doi: 10.1155/2012/971963. Epub 2012 Jun 25. PMID 22792099
- [Result] Chen HP, Shen SJ, Tsai HI, Kao SC, Yu HP. Effects of Interscalene Nerve Block for Postoperative Pain Management in Patients after Shoulder Surgery. Biomed Res Int. 2015;2015:902745. doi: 10.1155/2015/902745. Epub 2015 Nov 24. PMID 26688821
- [Result] Cabaton J, Nove-Josserand L, Mercadal L, Vaudelin T. Analgesic efficacy of ultrasound-guided interscalene block vs. supraclavicular block for ambulatory arthroscopic rotator cuff repair: A randomised noninferiority study. Eur J Anaesthesiol. 2019 Oct;36(10):778-786. doi: 10.1097/EJA.0000000000001065. PMID 31361631